CLINICAL TRIAL: NCT02996006
Title: New Techniques to Reduce Intra-operative Bleeding During Complex Liver Resection
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lei Dou, Registrar, Tongji Hospital
Other Study IDs: TJ-liver-200804
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Surgical Blood Loss
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

INTERVENTIONS:
Procedure: stepwise vascular control — Before liver parenchymal resection, we performed "total hepatic vascular preparation for occlusion" with portal triad (PT), infra-hepatic inferior vena cava (IIVC), and supra-hepatic inferior vena cava (SIVC) preparation in order. Then we performed step-by-step vascular occlusion according to the individual bleeding situation.

SUMMARY:
This observational study introduced an new advanced bleeding control strategy during complex liver resection.This newly described "stepwise vascular control" technique was efficacious and feasible to control intra-operative bleeding in complex hepatectomy involving second hepatic hilum and retro-hepatic inferior vena cava.

ELIGIBILITY:
Inclusion Criteria:

* tumor size is more than 5cm in diameter;
* these tumor were close to or were compressing main hepatic veins and RIVC directly;
* Pugh-Child Grade is A or Indocyanine green retention rate at 15min (ICG15%) is less than 10% .

Ages: 41 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patient sampling according to the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
blood loss during liver resection | duration of operation time

REFERENCES:
- [Derived] Dou L, Yu ZP, Yang HY, Ran J, Chen YF, Chen XP. Personalized stepwise vascular control during complex hepatectomy involving hepatocaval confluence. ANZ J Surg. 2018 Jul-Aug;88(7-8):E606-E609. doi: 10.1111/ans.14301. Epub 2017 Dec 10. PMID 29224239